CLINICAL TRIAL: NCT02818322
Title: The Role of Telemedical Monitoring in Diabetic Foot Ulcer Care
Acronym: A15-06
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PA15083
Record Dates: First submitted 2016-06-23; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Diabetic Foot - Telemedical Monitoring

ARMS (2):
- telemedical monitoring ( T) (Experimental): Home care by a nurse trained in the management of diabetic foot lesions with transmission diabetologist doctor a photograph and a full description of the diabetic foot lesion every week
  Interventions: Device: telemedical monitoring ( T); Device: classic monitoring
- classic monitoring (Active Comparator): Home care by a nurse trained in the management of diabetic foot lesions without transmission diabetologist doctor a photograph and a full description of the diabetic foot lesion
  Interventions: Device: classic monitoring

INTERVENTIONS:
Device: telemedical monitoring ( T)
  Arms: telemedical monitoring ( T)
Device: classic monitoring

SUMMARY:
The role of telemedical monitoring in diabetic foot care is still uncertain. The aim is to compare telemedical + standard and standard alone outpatient monitoring in the care of patients with diabetic foot ulcers in a randomized controlled trial. The primary outcome of the overall study is the time of ulcer healing. The number of amputation, hospital admissions and surgical procedure will be also reported. Investigators hope to include 150 patients in this study.

ELIGIBILITY:
Inclusion Criteria:

* The patients treated in the diabetology department of CHU de Reims during the inclusion phase to a diabetic foot lesions ( infected or not).
* Patients with care of this lesion of diabetic foot externally.
* Patients who agreed to participate in or accepting ORNICARE network ( network for the transmission of information between health care professionals) (Appendix 3) .
* Patients aged over 18 years .
* Patients who agreed to participate in the study .
* The patients insured by a social security scheme .

Exclusion Criteria:

* Patients requiring hospital care of the lesion of diabetic foot (infection requiring surgical intervention , ischemia requiring revascularization , ...).
* Patients are protected by law .
* Minor patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
time of ulcer healing | 6 month after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France